CLINICAL TRIAL: NCT00805402
Title: Interest of Flow Cytometry for the Diagnosis, the Follow up and SIT Arrest of Hymenoptera Venom Allergy
Brief Title: Interest of Flow Cytometry for the Diagnosis, the Follow up and Specific Immunotherapy (SIT) Arrest of Hymenoptera Venom Allergy
Acronym: Cytoven
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I07021
Record Dates: First submitted 2008-12-02; First posted 2008-12-09 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2010-09

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 flow cytometry (Experimental): flow cytometry
  Interventions: Other: flow cytometry

INTERVENTIONS:
Other: flow cytometry — flow cytometry

SUMMARY:
The aim of this study is to show that flow cytometry can be an accurate tool to help physicians regarding the diagnosis, the SIT decision and the SIT arrest of hymenoptera venom allergy.

75 patients having a story of reaction to hymenoptera venom will be selected for this trial.

Blood samples will be analyzed at: inclusion visit, Week 1 visit, Week 3 visit, Week 10 and Week 21 visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18 - 70 years)
* Patient being informed and accepting to participate in the study with signature of informed consent
* Patients having a clinical systematic and local, loco-regional story of reaction to the piqures of hymenopterans.
* Patients treated by SIT for at least 5 years
* Patients benefiting from a national insurance health

Exclusion Criteria:

* Children
* Pregnant woman or who breast-feed
* Patient under antihistaminic or corticoid for less than 8 days before the blood drawing
* Protected Patient
* Patient not having given his agreement after it was informed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
% CD63 expression on basophil membrane by flow Cytometry | Inclusion , Week 1, Week 3, Week 10 and Week 21 visits

SECONDARY OUTCOMES:
Blood blocking factors level | Week 1, Week 3, Week 10 and Week 21 visits

CONTACTS AND LOCATIONS:
Overall Officials: Michel COGNE, MD, Principal Investigator — CHU Limoges; Jean Sainte-Laudy, PhD, Study Chair — CHU Limoges
Locations (1):
- Service Pathologie Respiratoire, Limoges, France

REFERENCES:
- [Background] Sainte-Laudy J, Touraine F, Cluzan D, Belle Moudourou F. Follow-Up of Venom Immunotherapy on Flow Cytometry and Definition of a Protective Index. Int Arch Allergy Immunol. 2016;170(4):243-250. doi: 10.1159/000449162. Epub 2016 Sep 30. PMID 27685197